#### INFORMED CONSENT FORM

**September 24, 2025** 

# Research Project Title: The Effect of Wellness Coaching and Mobile Applications on Psychosocial Adjustment and Well-Being to Women Newly Diagnosed with Breast Cancer

You have been invited to participate in a study titled "The Effect of Wellness Coaching and Mobile Applications on Psychosocial Adjustment and Well-Being to Women Newly Diagnosed with Breast Cancer." You have been invited to participate because you have been diagnosed with breast cancer. This study is being conducted for research purposes, and participation is voluntary. Before you decide to participate, we would like to inform you about the study. After you have been fully informed about the study and your questions have been answered, you will be asked to sign this form if you wish to participate. This research is being conducted at the Medical Oncology Outpatient Clinic of SBU Gülhane Training and Research Hospital under the supervision of Prof. Dr. It is carried out by the researcher Gülhane Faculty of Nursing, Public Health Nursing Department Assoc. Prof. Dr. Şeyma Zehra ALTUNKÜREK and Specialist Nursing Assistant Eylül YEŞİLYURT, with the knowledge of Nuri KARADURMUŞ.

## What is the purpose of the study? How many people, in addition to me, will participate in this study?

The purpose of this study is to determine the effects of Mobile Wellness Coaching and Group Wellness Coaching programs on the psychosocial adjustment and well-being of women newly diagnosed with breast cancer. This study is being conducted for research purposes only.

The study is a single-center study conducted at the Medical Oncology Outpatient Clinic of SBU Gülhane Training and Research Hospital. The study is planned to include 124 people.

### Should I participate in this study?

Whether or not you choose to participate in this study is entirely up to you. Even if you sign this form now, you are free to withdraw at any time without giving a reason.

### What will happen if I participate in this study?

If you participate in the study, you are expected to participate in the training programs developed by the researchers and use the mobile app. Wellness Coaching programs designed for women diagnosed with breast cancer will be delivered via the mobile app and in groups. The program content is designed to facilitate your adjustment to the disease and enhance your well-being. The researchers have completed their coaching training through certification programs and are experts in their field.

If you agree to participate in the study, you will be asked to complete a survey. This form was developed

by the researchers and consists of "Descriptive Information," "Information About the Illness,"

"Psychosocial Adjustment to the Illness-Self-Report Scale (PAIS-SR)," and "Holistic Well-Being Scale."

You will then be expected to attend a total of eight wellness coaching trainings, one day per week for

eight weeks. You will also be able to access the wellness training through the mobile app. Each training

session is planned to last 45-50 minutes. You will be asked to complete a survey immediately after the

training, one month later, and three months later. The survey form, consisting of the "Psychosocial

Adjustment to the Illness-Self-Report Scale (PAIS-SR)" and the "Holistic Well-Being Scale," will be sent

to you as a Google Survey form. This will complete the study.

Are there any risks or discomforts associated with the study?

All expenses related to the study will be covered by us. The study poses no risks or discomforts for you.

What are the benefits of participating in the study?

In women newly diagnosed with breast cancer, helping them adapt to the disease and improving their

well-being allows them to respond more quickly to treatment. In this case, the wellness coaching training

we will provide you with will help you better manage this process.

What is the cost of participating in this study?

You will not be financially burdened by participating in the study, and no payment will be made to you.

The Social Security Institution (SGK) will not be billed.

How will my personal information be used?

Your personal information will not be collected as part of the study. Your contact number will be required

to contact you and schedule groups. Your responses to the survey questions will be used by the

researchers to conduct the study and statistical analyses. Ethics committees or official authorities may

review your information only if necessary. At the end of the study, you have the right to request

information about your results. The study results may be published in the medical literature upon

completion, but your identity will not be disclosed.

Who can I contact for more information?

If you need additional information about the study, please contact the person below.

NAME: Eylül YEŞİLYURT

POSITION: Specialist Nurse

PHONE: +905061108000

(Declaration of Participant/Patient)

I was informed that a study would be conducted by Associate Professor Dr. Şeyma Zehra ALTUNKÜREK and Specialist Eylül YEŞİLYURT at the Medical Oncology Outpatient Clinic of SBÜ Gülhane Training and Research Hospital, and the above-mentioned information about this study was provided to me, and I read the relevant text. Following this information, I was invited to participate as a "participant" in this research.

I have not been subjected to any coercive behavior regarding my participation in the research. I understand that there will be no harm if I refuse to participate. I may withdraw from the research without giving any reason during the project's implementation. (However, I am aware that it would be appropriate to notify the researchers in advance of my withdrawal to avoid putting them in a difficult situation.)

I assume no financial responsibility for any expenses incurred in the research, and no payment will be made to me.

I understand that the confidentiality of personal information obtained from the research will be protected.

I have fully understood all the explanations given to me. Under these conditions, I agree to participate in this research voluntarily, without any pressure or coercion. A copy of this signed form will be given to me.

| Participant (Handwritten) |
|---------------------------|
| Name, surname: |
| Address: |
| Phone: |
| Signature: |
| Date: |
| Researcher (Handwritten) |
| Name, surname, title: |
| Address: |
| Phone: |
| Signature: |

Date: